CLINICAL TRIAL: NCT00127491
Title: A RCT of Mechanical Ventilation, Directed by Esophageal Pressure Measurements, in Patients With Acute Lung Injury
Brief Title: Mechanical Ventilation, Directed by Esophageal Pressure Measurements, in Patients With Acute Lung Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Talmor, Edward Lowenstein Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004P000011; R01HL052586 (NIH)
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Mechanical Ventilation; Esophageal Pressures; Randomized Controlled Trial
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPVent (Experimental): All patients will have an esophageal balloon placed for the purpose of obtaining transpulmonary pressure measurements. The intervention group will undergo transpulmonary pressure-directed controlled mechanical ventilation using parameters directed by the initial balloon measurements. Driving pressures will be adjusted to maintain a transpulmonary plateau pressure of less then 30. The PEEP setting will be set to achieve a transpulmonary end expiratory pressure of 0. Repeat PES measurements will be done at 24, 48 and 72 hours following the initial measurements. Additional measurements will be taken as clinically indicated. Ventilator management by PES measurements will continue for a period of 72 hours.
  Interventions: Procedure: Placement of an esophageal balloon measurements; Other: Transpulmonary pressure-directed ventilation (EPVent)
- Control (Active Comparator): All patients will have an esophageal balloon placed for the purpose of obtaining transpulmonary pressure measurements. The control group will be managed using the low tidal volume strategy laid out by the NIHBLI ARDSnet study. These recommendations include a set tidal volume of 6 ml/ kg. Respiratory rate and PEEP are set to maintain adequate ventilation and oxygenation. These settings will be continued for a period of 72 hours.
  Interventions: Procedure: Placement of an esophageal balloon measurements; Other: Low tidal volume ventilation

INTERVENTIONS:
Procedure: Placement of an esophageal balloon measurements — In both groups an esophageal balloon will be placed and baseline measurements recorded. In the EP group the mechanical ventilation settings will be determined based on these measurements. In the control group measurements will be recorded but ventilation will be based in the existing standard of care wich is the ARDSnet low tidal volume ventilation study. measurements will be repeated at 24, 48 and 72 hours or as needed.
Other: Low tidal volume ventilation — Low tidal volume ventilation strategy (ARDSnet)
  Arms: Control
Other: Transpulmonary pressure-directed ventilation (EPVent) — Transpulmonary pressure-directed ventilation using measurements from the esophageal balloon.
  Arms: EPVent

SUMMARY:
The purpose of this study is to see whether esophageal pressure (PES) measurements will allow the investigators to choose the best method of mechanical ventilation in patients with acute lung injury (ALI).

DETAILED DESCRIPTION:
The current standard of practice for ventilating patients with acute respiratory distress syndrome (ARDS) is the ARDSnet protocol (N Engl J Med 2000; 342:1301-1308) which has been shown to improve survival by limiting tidal volumes and thus preventing over distention of the lungs. However, the lungs can also be damaged by under-inflation during mechanical ventilation, and current practice ignores the effects of chest wall compression of the lungs, which can cause under-inflation. The investigators have observed that a fraction of critically ill patients with apparent ARDS have lung function abnormalities caused by extrinsic compression which can be estimated by PES measurements. Changing ventilator settings to apply normal physiological pressure to the lung has been beneficial in many such patients. This protocol will formally test the clinical utility of PES measurements in patients with ARDS.

This is a randomized controlled trial of therapy directed by esophageal balloon measurements (PES) versus therapy directed by ARDSnet protocol, the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

Patients with ALI/ARDS according to the International Consensus Conference criteria:

* PaO2/FiO2 ratio < 300
* Acute onset
* Bilateral infiltrates on chest radiography
* PAOP < 18 or, in patients without a pulmonary artery catheter, no other evidence of abnormal cardiac function

Exclusion Criteria:

* Patients with esophageal varices
* Patients with esophageal trauma
* Patients with recent esophageal surgery
* Patients with coagulopathy (platelets < 80k or International Normalized Ratio [INR]> 2 )
* Post transplant patients
* Patients with significant broncho-pleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-05; Primary Completion 2007-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Oxygenation as measured by the PO2/FiO2 (P/F) ratio | 72 hours from enrollment

SECONDARY OUTCOMES:
Ventilator free days | At 28 days
Markers of inflammation | In first 72 hours
Mortality | At 28, 90 and 180 days
Length of stay | Hospital and ICU

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Talmor, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loring SH, O'Donnell CR, Behazin N, Malhotra A, Sarge T, Ritz R, Novack V, Talmor D. Esophageal pressures in acute lung injury: do they represent artifact or useful information about transpulmonary pressure, chest wall mechanics, and lung stress? J Appl Physiol (1985). 2010 Mar;108(3):515-22. doi: 10.1152/japplphysiol.00835.2009. Epub 2009 Dec 17. PMID 20019160
- [Background] Sarge T, Talmor D. Targeting transpulmonary pressure to prevent ventilator induced lung injury. Minerva Anestesiol. 2009 May;75(5):293-9. PMID 19412147
- [Result] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Derived] Schaefer MS, Loring SH, Talmor D, Baedorf-Kassis EN. Comparison of mechanical power estimations in mechanically ventilated patients with ARDS: a secondary data analysis from the EPVent study. Intensive Care Med. 2021 Jan;47(1):130-132. doi: 10.1007/s00134-020-06282-1. Epub 2020 Oct 19. No abstract available. PMID 33078240
- [Derived] Talmor D, Sarge T, Legedza A, O'Donnell CR, Ritz R, Loring SH, Malhotra A. Cytokine release following recruitment maneuvers. Chest. 2007 Nov;132(5):1434-9. doi: 10.1378/chest.07-1551. Epub 2007 Oct 9. PMID 17925413